CLINICAL TRIAL: NCT05743985
Title: Efficacy and Safety of Hemp-derived, Full Spectrum Cannabigerol (CBG) in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Formula30A LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F30A-CBG-EAS2022
Record Dates: First submitted 2023-02-15; First posted 2023-02-24 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Health, Subjective; Inflammatory Response; Adverse Effect; Side Effect
Keywords: Endocannabinoid System; Cannabis; Cannabigerol; CBG; Cannabinoids; Cannabinoid; Hemp
MeSH Terms: conditions — Marijuana Abuse | interventions — cannabigerol; Calcium Gluconate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 50mg CBG Capsule (Experimental): 50mg cannabigerol (CBG) oil capsule taken daily for 8 weeks. Study surveys and bloodwork completed for 12 weeks total, including 8 weeks of CBG treatment and subsequent 4-week washout period
  Interventions: Other: Cannabigerol

INTERVENTIONS:
Other: Cannabigerol — Hemp-derived full spectrum cannabigerol oil carried in an organic coconut (MCT) oil within hydroxypropyl methylcellulose capsules.
  Other Names: Formula30A Cannabigerol (CBG) 50mg Capsules; Formula30A CBG

SUMMARY:
The goal of this observational study is to provide exploratory research into the in vivo physiological and psychological effects, if any, of cannabigerol (CBG) in healthy human adults age 21 or over.

The main questions it aims to answer are:

* What effect, if any, does daily oral consumption of 50mg of full spectrum CBG have on the mental, physical, and emotional wellbeing of healthy individuals, as measured by self-report Medical Symptom Questionnaire and 36-Item Short Form Health Survey scores?
* Is CBG effective at reducing inflammation in the body, as measured by HSCRP, ESR, and PSA inflammatory markers?
* Do age, gender, weight, or state of body inflammation have an effect on the perceived efficacy of CBG?
* What adverse effects, if any, are associated with CBG use?

Over the course of the 12-week study, participants will:

* Take baseline MSQ and SF-36 surveys, as well as a clinical visit with blood draws for HSCRP, ESR, and PSA testing
* Consume one (1) 50mg capsule of full spectrum CBG daily by mouth with food for 8 weeks, followed by a 4-week washout period
* Complete biweekly SF-36 surveys as well as MSQ surveys every 4 weeks
* Attend a clinical visit every 4 weeks for clinical observation and blood draws for HSCRP, ESR, and PSA (male subjects)

DETAILED DESCRIPTION:
BACKGROUND AND CONTEXT

The Cannabis plant has gained significant, and increasing, interest in the medical community due to the therapeutic potential of substances such as Δ9-tetrahydrocannabinol (Δ9-THC) and cannabidiol (CBD). However, there are hundreds of different phytocannabinoids, terpenes, and flavonoids present in Cannabis plants, generating complex interactions in the human body. Cannabigerol (CBG) is one phytocannabinoid that has recently garnered a groundswell of media and commercial interest, although scientific literature on CBG is severely lacking compared with published research on Δ9-THC and CBD. Current studies suggest that CBG appears to have characteristics for affinity and activity somewhere between CBD and Δ9-THC, with additional unique interactions with 5-hydroxytryptamine (5-HT1A) receptors and α-2 adrenoceptors. Based on published research, there may be therapeutic potential for CBG in the treatment of neuroinflammatory disorders, inflammatory bowel disease, bacterial infections (such as MRSA), prostate cancer, and dental plaque. Many of these studies, however, indicate a vital need for additional research on the pharmacological effects of human CBG consumption, especially given the increase in its unregulated commercial use. This study will focus on the clinical application of CBG for healthy adults, current knowledge of its possible therapeutic utility, and its potential toxicological hazards.

PROBLEM STATEMENT

Cannabigerol is currently available for purchase in a variety of products and, as with cannabidiol (CBD) before it, many claims are being made about its benefits. Unlike CBD, however, little in-depth research has been performed on this intriguing phytocannabinoid, and much of what is known warrants further investigation to identify potential areas of therapeutic uses and hazards.

RESEARCH QUESTIONS

What effect, if any, does daily oral consumption of 50mg of full spectrum CBG have on the mental, physical, and emotional wellbeing of healthy individuals, as measured by self-report Medical Symptom Questionnaire and 36-Item Short Form Health Survey scores? Is CBG effective at reducing inflammation in the body, as measured by HSCRP, ESR, and PSA inflammatory markers? Do age, gender, weight, or state of body inflammation have an effect on the perceived efficacy of CBG? What adverse effects, if any, are associated with CBG use?

OBJECTIVES

The long-term goal is to provide exploratory research into the in vivo physiological and psychological effects, if any, of cannabigerol in humans. The objective of the current study is to determine whether clinically applied CBG in 100 healthy adults 21 or over in the United States has an effect on inflammatory markers in the body and/or self-reported physical, mental, and emotional wellbeing. The study has the following sub-objectives:

1. To provide initial data on the physiological and self-reported psychological effects CBG;
2. To work towards development of a CBG administration method for easier physician dosage control and oversight;
3. To review and document current industry practices and research in regard to CBG use;
4. To outline a conceptual framework for the clinical application of CBG.

The result of this study will be valuable to industry practitioners as well as patient populations in developing a clear pharmacological picture of the efficacy and risks of full spectrum CBG consumption.

ELIGIBILITY:
Inclusion Criteria:

* In good overall health (as determined by the supervising healthcare provider recommendation as well as no indications of Moderate or Severe conditions on the study measurement tools)
* 21 years old or over
* No conditions determined at risk for adverse reactions to the product ingredients
* Research participants with the potential to become pregnant are eligible to be included in the study as long as they are sexually abstinent or using a contraceptive method considered effective.

Exclusion Criteria:

* Under the age of 21
* Is pregnant or breastfeeding
* Initiated or changed use of medication or therapies within 2 weeks prior to the start of the study
* Has a history of hepatic compromise (with transaminases of two times the upper limit of normal) or cirrhosis
* Is already using recreational marijuana, medical marijuana or other cannabinoid formulations (including CBD)
* Has a history of substance or alcohol abuse
* Is using High Dose or Extended-Release Narcotics

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Medical Symptom Questionnaire (MSQ) Score at 8 weeks | 8 weeks
  Change from baseline scores as measured by the Medical Symptom Questionnaire after 8 weeks. A total score of 20 or less is not clinically significant, 20 to 49 indicates mild toxicity, 50 to 99 indicates moderate toxicity, and 100 and above indicates severe toxicity.
Change from Baseline RAND 36-Item Short Form Survey (SF-36) Scores at 8 weeks | 8 weeks
  Change from baseline scores as measured by the RAND 36-Item Short Form Survey after 8 weeks. Scores range from 0-100 for the 8 scales included (physical functioning, role limitations due to physical health, role limitations due to emotional problems, energy/fatigue, emotional well-being, social functioning, pain, and general health), with higher scores representing a more favorable health state.
Change from Baseline High-Sensitivity C-reactive Protein (hsCRP) at 8 weeks | 8 weeks
  Blood concentration, measured in mg/L
Change from Baseline Erythrocyte Sedimentation Rate (ESR) at 8 weeks | 8 weeks
  Blood concentration, measured in mm/hour
Change from Baseline Prostate-Specific Antigen (PSA) Score at 8 weeks [Male Subjects] | 8 weeks
  Blood concentration, measured in ng/mL

CONTACTS AND LOCATIONS:
Overall Officials: Cory Rice, D.O., Principal Investigator — Modern Medicine
Locations (6):
- United States (5):
  - Institute for Hormonal Balance, Arlington, Texas
  - NP Care Clinic, Denton, Texas
  - Infectious Disease Specialists, Edinburg, Texas
  - Modern Medicine, Forney, Texas
  - Melville Medicine, Southlake, Texas
- Java Med, Ceiba, Puerto Rico, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication, shared upon request.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Starting 6 months after publication.
Access Criteria: IPD and additional supporting information shared upon request.

REFERENCES:
- [Background] Nachnani R, Raup-Konsavage WM, Vrana KE. The Pharmacological Case for Cannabigerol. J Pharmacol Exp Ther. 2021 Feb;376(2):204-212. doi: 10.1124/jpet.120.000340. Epub 2020 Nov 9. PMID 33168643
- [Background] Navarro G, Varani K, Reyes-Resina I, Sanchez de Medina V, Rivas-Santisteban R, Sanchez-Carnerero Callado C, Vincenzi F, Casano S, Ferreiro-Vera C, Canela EI, Borea PA, Nadal X, Franco R. Cannabigerol Action at Cannabinoid CB1 and CB2 Receptors and at CB1-CB2 Heteroreceptor Complexes. Front Pharmacol. 2018 Jun 21;9:632. doi: 10.3389/fphar.2018.00632. eCollection 2018. PMID 29977202
- [Background] De Petrocellis L, Ligresti A, Moriello AS, Allara M, Bisogno T, Petrosino S, Stott CG, Di Marzo V. Effects of cannabinoids and cannabinoid-enriched Cannabis extracts on TRP channels and endocannabinoid metabolic enzymes. Br J Pharmacol. 2011 Aug;163(7):1479-94. doi: 10.1111/j.1476-5381.2010.01166.x. PMID 21175579
- [Background] Echeverry C, Prunell G, Narbondo C, de Medina VS, Nadal X, Reyes-Parada M, Scorza C. A Comparative In Vitro Study of the Neuroprotective Effect Induced by Cannabidiol, Cannabigerol, and Their Respective Acid Forms: Relevance of the 5-HT1A Receptors. Neurotox Res. 2021 Apr;39(2):335-348. doi: 10.1007/s12640-020-00277-y. Epub 2020 Sep 4. PMID 32886342
- [Background] Fellous T, De Maio F, Kalkan H, Carannante B, Boccella S, Petrosino S, Maione S, Di Marzo V, Iannotti FA. Phytocannabinoids promote viability and functional adipogenesis of bone marrow-derived mesenchymal stem cells through different molecular targets. Biochem Pharmacol. 2020 May;175:113859. doi: 10.1016/j.bcp.2020.113859. Epub 2020 Feb 14. PMID 32061773
- [Background] Crocq MA. History of cannabis and the endocannabinoid system . Dialogues Clin Neurosci. 2020 Sep;22(3):223-228. doi: 10.31887/DCNS.2020.22.3/mcrocq. PMID 33162765
- [Background] Russo EB, Cuttler C, Cooper ZD, Stueber A, Whiteley VL, Sexton M. Survey of Patients Employing Cannabigerol-Predominant Cannabis Preparations: Perceived Medical Effects, Adverse Events, and Withdrawal Symptoms. Cannabis Cannabinoid Res. 2022 Oct;7(5):706-716. doi: 10.1089/can.2021.0058. Epub 2021 Sep 27. PMID 34569849